CLINICAL TRIAL: NCT06756308
Title: A Phase 2 Study of Enasidenib in IDH2-Mutant Angioimmunoblastic T-Cell Lymphoma
Brief Title: A Study of Enasidenib in People With T-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-269
Record Dates: First submitted 2024-12-27; First posted 2025-01-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: T-cell Lymphoma
Keywords: Enasidenib; Rituximab; IDH2-mutant; 23-269
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — enasidenib; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enasidenib and rituximab (Experimental): Screening Cohort (Non-MSK Patients only) Non-MSK patients will send research tissue samples to MSK for ddPCR analysis to assess IDH2 mutation. Once mutation is confirmed they may be consented to the treatment portion of the trial.
  All patients will receive oral enasidenib 100 mg daily on 28-day cycles. Patients with evidence of a co-occurring B-cell lymphoproliferation (via tumor morphology, flow cytometry, or B-cell clonality) will be administered IV rituximab 375 mg/m² weekly for the first month, and monthly for 3 months thereafter on 28-day cycles, for a total of four months of rituximab. If B-cell proliferation persists at the end of the 4-month rituximab treatment period, continue treatment with monthly rituximab until no evidence of B-cell lymphoproliferation is seen.
  Interventions: Drug: Enasidenib; Drug: Rituximab

INTERVENTIONS:
Drug: Enasidenib — Enasidenib 100 mg daily on 28-day cycles.
Drug: Rituximab — IV rituximab 375 mg/m² weekly for the first month, and monthly thereafter on 28-day cycles, for a total of four months of rituximab.

SUMMARY:
The researchers are doing this study to find out whether enasidenib is a safe treatment for people with angioimmunoblastic T-cell lymphoma (AITL) that has an IDH2 mutation. The researchers will look at the safety of enasidenib when it is given alone or in combination with the drug rituximab.

ELIGIBILITY:
Inclusion Criteria:

Screening Cohort (non-MSK patients only)

1. Age ≥18 years at time of consent
2. Has freely given written informed consent to participate in the study

Treatment Cohort:

1. Pathologically-confirmed AITL at the enrolling institution, with confirmed IDH2 mutation (by MSK ddPCR). For R/R patients, disease must have relapsed or progressed after at least one systemic therapy, diagnostic tumor samples have at least 5% tumor.
2. Age ≥18 years at time of enrollment
3. Previous systemic anti-cancer therapy for AITL must have been discontinued at least 2 weeks or 5 half-lives (whichever is longer) prior to treatment.

   i) See section 6.2 Subject Exclusion Criteria for guidelines regarding adjuvant and maintenance therapy for prior malignancy.

   ii) Patients who have received localized RT as part of their immediate prior therapy may be allowed to enroll with shorter washout period after discussion with the MSKCC Principal Investigator iii) Systemic corticosteroids must be tapered to 25 mg/day prednisone (or equivalent) upon start of investigational treatment iv) Topical steroids for treating cutaneous involvement of AITL is permitted
4. Performance status, as assessed in the ECOG grading system, ≤2
5. Laboratory criteria (use of GCSF and/or blood product transfusions to reach eligibility criteria must be discussed with the MSK PI on a case-by-case basis): i) Absolute neutrophil count ≥1.0 K/μL or ≥0.5 K/μL if due to lymphoma ii) Platelet count ≥80 K/μl or ≥50 K/μl if due to lymphoma iii) Calculated creatinine clearance ≥30 mL/min by the Modification of Diet in Renal Disease (MDRD) glomerular filtration rate iv) Total bilirubin ≤1.5x upper limit of normal (ULN) or ≤3x ULN if documented hepatic involvement with lymphoma, or ≤5x ULN if history of Gilbert's syndrome; AST and ALT ≤ 3x ULN; ≤ 5x ULN if due to lymphoma involvement
6. Measurable disease, defined by either of:

   * Revised International Working Group Classification for systemic lymphoma(13)
   * Atypical T lymphocytes quantifiable by flow cytometry or morphology in the peripheral blood or bone marrow
7. Women of reproductive potential* must have a negative serum or urine β human chorionic gonadotropin (β-hCG) pregnancy test. All women of reproductive potential must agree to use adequate methods of birth control throughout the study and for 30 days after the last dose of study drug. *A woman of reproductive potential is a sexually mature woman who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
8. Women must agree to not breastfeed during the study period
9. Male subjects must agree to practice true abstinence from sexual intercourse or to the use of highly effective contraceptive methods with non-pregnant female partners of childbearing potential at screening and throughout the course of the study, and should avoid conception with their partners during the course of the study and for 4 months following the last study treatment
10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. On immunosuppressive therapy post-allogeneic stem cell transplantation at the time of screening, or with clinically significant graft-versus-host disease (GVHD). The use of a stable dose of oral steroid post-HSCT and/or topical steroids for ongoing skin GVHD is permitted after discussion with the study PI
3. Subject has persistent, clinically significant non-hematologic toxicities grade >1 or not to baseline level from prior therapies besides alopecia or neuropathy
4. Pregnant women
5. History of chronic liver disease, veno-occlusive disease, or alcohol abuse
6. Administration of a live vaccine within 6 weeks of first dose of study drug
7. Prior surgery or gastrointestinal condition that may adversely affect drug absorption (e.g.,gastric bypass surgery, gastrectomy)
8. Patients with HIV infection with detectable viral load, CD4 count <200, or not taking anti-retroviral medications
9. Patients with chronic hepatitis B or C as defined by positive hepatitis B or C serology:

   1. Subjects with a negative HBsAg and a positive HBcAb require an undetectable/negative hepatitis B DNA test (e.g., polymerase chain reaction [PCR] test) to be enrolled, and will require prophylactic antiviral treatment according to institutional standards of care initiated prior to the first dose of study drug, and continued until approximately 18 months after completion of study drug(s) if rituximab is utilized.
   2. Patients who are hepatitis C antibody positive with negative PCR may enroll
10. Subjects with active CMV (defined as positive serum CMV PCR with clinical manifestations consistent with active CMV infection) and requiring therapy. Carriers (low-level positivity by PCR and without evidence of CMV disease) will be monitored per institutional guidelines when such guidelines exist or individual physician practice in the absence of formal guidelines to ensure stability in the PCR level over time and continued absence of CMV disease manifestations.
11. Receiving therapy for another primary malignancy (other than T-cell lymphoma).

    1. Patients with more than one type of lymphoma may be enrolled after discussion with the MSK Principal Investigator.
    2. Early-stage cutaneous basal cell and squamous cell carcinomas are permissible
    3. Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy is potentially permissible after discussion with the MSK Principal Investigator.
12. Known central nervous system or meningeal involvement by AITL (in the absence symptoms, investigation into central nervous system involvement is not required)
13. Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
14. Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to the start of study treatment.
15. Prior use of enasidenib
16. Subjects taking the following sensitive CYP substrate medications with narrow therapeutic ranges are excluded from enrolment the study unless they can be safely rotated to other medications within >4 half-lives prior to C1D1: warfarin and phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline and tizanidine (CYP1A2).
17. Subjects taking the P-gp- and BCRP transporter-sensitive substrates digoxin and rosuvastatin should be counseled with pharmacy input regarding drug-drug interactions.

    1. Digoxin is acceptable with dose modification after consulting with a pharmacist
    2. Patients taking rosuvastatin should be excluded from the study unless they can safely be rotated to alternative medications within >4 half-lives prior to C1D1.
18. Caution should be exercised on patients on medications that are substrates for UGT1A1 (including but not limited to ezetimibe, raloxifene, and raltegravir). Such patients shall rotate to alternate therapies, or reduce doses of these medications in consultation with the prescribing provider and/or a consulting pharmacist. Close monitoring for adverse events shall be pursued in these instances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
response rate | 1 year
  a 20% response rate is undesirable and 45% is desirable

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Epstein-Peterson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Dana Farber Cancer Institute (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm